CLINICAL TRIAL: NCT03413514
Title: A Non-Randomized,Single Center Study to Investigate the Real World Evidence for the Maximal Cycle of Effective Neoadjuvant Chemotherapy in Gastric Cancer With Shared Decision Making
Brief Title: Real World Evidence for the Cycle of Neoadjuvant Chemotherapy in Gastric Cancer With Shared Decision Making
Acronym: RECOMMEND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, Chief Physician, Professor, Peking University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017YJZ51
Record Dates: First submitted 2018-01-14; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
Keywords: shared decision making; neoadjuvant chemotherapy; cycle; MRI; clinical response
MeSH Terms: conditions — Stomach Neoplasms | interventions — SDM; Surgical Procedures, Operative; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment group (Experimental): Neoadjuvant chemotherapy(NACT) are performed for locally advanced gastric cancer. The clinical response is evaluated by MRI and enhanced CT. The cycle of neoadjuvant chemotherapy is decided by the doctor and the patents together with shared decision making(SDM). Radical gastrectomy with D2 lymph node dissection are performed after neoadjuvant chemotherapy. Adjuvant chemotherapy(ACT) are preformed after surgery. Questionnaires are preformed to evaluate the involvement emotion and reason for the decision of stopping neoadjuvant chemotherapy.
  Interventions: Drug: NACT; Procedure: SDM; Procedure: Surgery; Drug: ACT; Other: Questionnaire

INTERVENTIONS:
Drug: NACT — SOX: Oxaliplatin 130mg/m2,iv.,d1; S-1 60mg,po.,Bid,d1-14; Repeat every 21 days for n courses.(0<n<8)
Procedure: SDM — Making the decision about the cycle of neoadjuvant chemotherapy with shared decision making
Procedure: Surgery — Radical surgery with D2 lymph node dissection
Drug: ACT — SOX: Oxaliplatin 130mg/m2,iv.,d1; S-1 60mg,po.,Bid,d1-14; Repeat every 21 days for 8-n courses.(0<n<8)
Other: Questionnaire — MAPPIN'SDM questionnaire, the control performance card, the care questionnaire, the decisional conflict questionnaire, the decisional regret questionnaire, the questionnaire of the reason for stopping neoadjuvant chemotherapy

SUMMARY:
The purpose of the study is to evaluate the maximal cycle of effective neoadjuvant chemotherapy for resectable gastric cancer, to determine what is the best cycle of neoadjuvant chemotherapy for the patients who receive neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The study is a non-randomized clinical trial. The protocol has been approved by the Ethics Committee of Beijing Cancer Hospital. MRI and enhanced CT are used to evaluate the clinical response of the tumor. The primary endpoint is the maximal cycle of effective neoadjuvant chemotherapy for resectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the stomach
2. Clinical cT2N+M0,or cT3-4a/N+M0 disease, confirmed by upper gastrointestinal endoscopy and abdominal computed tomography (CT) and MRI and laparoscopy.
3. Receive neoadjuvant chemotherapy in clinical

Exclusion Criteria:

1. Contraindication for chemotherapy
2. Contraindication for surgery
3. Clinically apparent distant metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-01-03 (Estimated); Study Completion 2023-01-03 (Estimated)

PRIMARY OUTCOMES:
The cycle of neoadjuvant chemotherapy | 18months
  The cycle of neoadjuvant chemotherapy means the maximal cycle of effective neoadjuvant chemotherapy. The effective means no disease progress by image diagnosis

SECONDARY OUTCOMES:
The clinical response rate | 18 months
  The clinical response is evaluated by CT/MRI according to the Response Evaluation Criteria In Solid Tumors (RECIST)1.1
The completion rate of perioperative chemotherapy | 18 months
  The completion rate of perioperative chemotherapy means the patient completed the 8 cycles of perioperative chemotherapy as planned (n cycles of neoadjuvant chemotherapy and 8-n cycles of adjuvant chemotherapy)
The progressive disease rate | 18 months
  The progressive disease during neoadjuvant chemotherapy with shared decision making is is evaluated by CT/MRI according to the Response Evaluation Criteria In Solid Tumors (RECIST)1.1
The pathological response | 18 months
  The pathological response during neoadjuvant chemotherapy with shared decision making is evaluated according to the tumor regression grade of NCCN guideline.
The pathological complete response | 18months
  The pathological complete response is defined as ypT0N0M0
The adverse event of chemotherapy | 18 months
  The adverse event of chemotherapy is evaluated and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) v.3
Surgical morbidity | 18 months
  Surgical morbidity is defined as the events which occurs with-in postoperative 30 days, extension of hospitalization and re-hospitalization. It is necessary to evaluate the complication and if it occurs during the hospitalization, it is required to record complication name, date of on-set (postoperatively), grade on Clavien-Dindo Classification and treatment for complication.
The 3-year progression-free survival | 48months
  In terms of locally advanced gastric cancer, to evaluate the progression-free survival rate in gastrectomy with D2 lymph node dissection at postoperative 3 years
The cTNM,ycTNM,ypTNM stage | 60months
  The cTNM stage, ycTNM stage and ypTNM stage is defined according to the 8th TNM stage.
The decisional conflicts | 12months
  The decisional conflicts is evaluated by Decisional Conflict Scale
The decisional regrets | 12months
  The decisional regrets is evaluated by Decision Regret Scale
The involvement of patients during the shared decision making | 12months
  The involvement of patients during the shared decision making is evaluated by MAPPIN'SDM questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Jiafu Ji, MD,PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Yoshikawa T, Tanabe K, Nishikawa K, Ito Y, Matsui T, Kimura Y, Hirabayashi N, Mikata S, Iwahashi M, Fukushima R, Takiguchi N, Miyashiro I, Morita S, Miyashita Y, Tsuburaya A, Sakamoto J. Induction of a pathological complete response by four courses of neoadjuvant chemotherapy for gastric cancer: early results of the randomized phase II COMPASS trial. Ann Surg Oncol. 2014 Jan;21(1):213-9. doi: 10.1245/s10434-013-3055-x. Epub 2013 Jul 10. PMID 23838904
- [Background] Aoyama T, Nishikawa K, Fujitani K, Tanabe K, Ito S, Matsui T, Miki A, Nemoto H, Sakamaki K, Fukunaga T, Kimura Y, Hirabayashi N, Yoshikawa T. Early results of a randomized two-by-two factorial phase II trial comparing neoadjuvant chemotherapy with two and four courses of cisplatin/S-1 and docetaxel/cisplatin/S-1 as neoadjuvant chemotherapy for locally advanced gastric cancer. Ann Oncol. 2017 Aug 1;28(8):1876-1881. doi: 10.1093/annonc/mdx236. PMID 28486692
- [Background] Schulz C, Kullmann F, Kunzmann V, Fuchs M, Geissler M, Vehling-Kaiser U, Stauder H, Wein A, Al-Batran SE, Kubin T, Schafer C, Stintzing S, Giessen C, Modest DP, Ridwelski K, Heinemann V. NeoFLOT: Multicenter phase II study of perioperative chemotherapy in resectable adenocarcinoma of the gastroesophageal junction or gastric adenocarcinoma-Very good response predominantly in patients with intestinal type tumors. Int J Cancer. 2015 Aug 1;137(3):678-85. doi: 10.1002/ijc.29403. Epub 2015 Feb 25. PMID 25530271
- [Background] Kane HL, Halpern MT, Squiers LB, Treiman KA, McCormack LA. Implementing and evaluating shared decision making in oncology practice. CA Cancer J Clin. 2014 Nov-Dec;64(6):377-88. doi: 10.3322/caac.21245. Epub 2014 Sep 8. PMID 25200391
- [Background] Fried TR. Shared Decision Making--Finding the Sweet Spot. N Engl J Med. 2016 Jan 14;374(2):104-6. doi: 10.1056/NEJMp1510020. No abstract available. PMID 26760081